CLINICAL TRIAL: NCT02187549
Title: Safety and Effectiveness Study of a Non-Crosslinked HA Alkylamide HYADD(TM) 4 Hydrogel for Osteoarthritis of the Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EQE7-13-01
Record Dates: First submitted 2014-06-29; First posted 2014-07-11 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Knee Osteoarthritis
Keywords: Hyaluronic Acid; Osteoarthritis; Knee; Hyaluronan; Viscoelastic; Hydrogel
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HYMOVIS (Experimental): HYADD(TM) 4 Hydrogel Intra-Articular Injection
  Interventions: Device: HYMOVIS
- Placebo (Placebo Comparator): Saline Intra-Articular Injection
  Interventions: Device: Placebo

INTERVENTIONS:
Device: HYMOVIS — Intra-articular injection
  Other Names: HYADD(TM) 4 Hydrogel Intra-Articular Injection
  Arms: HYMOVIS
Device: Placebo — Intra-Articular Injection
  Other Names: Placebo Intra-Articular Injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether intra-articular hyaluronic acid provides symptomatic relief of osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the knee.

Exclusion Criteria:

* No disorders which could interfere with study required assessments.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Pain Sub-score | 26 weeks

SECONDARY OUTCOMES:
Patient Global Assessment | 26 weeks

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Achieve Clinical Research, Birmingham, Alabama
  - Alabama Clinical Therapeutics, Brimingham, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Med Center, Carmichael, California
  - Triwest Research Associates, El Cajon, California
  - Westlake Medical, Thousand Oaks, California
  - Colorado Orthopedic Consultants, Englewood, Colorado
  - Chase Medical, Waterbury, Connecticut
  - Riverside Clinical Research, Edgewater, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Ormond Medical Arts, Ormond Beach, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Great Lakes Research Group, Bay City, Michigan
  - Healthcare Research Network, Hazelwood, Missouri
  - Fabio Orozco, Egg Harbor, New Jersey
  - PMG Research of Raleigh, Raleigh, North Carolina
  - New Horizons, Cincinnati, Ohio
  - Columbus Clinical Research, Columbus, Ohio
  - Blair Orphopedics, Altoona, Pennsylvania
  - West Houston Clinical Research, Houston, Texas